CLINICAL TRIAL: NCT03899714
Title: Return to Physical Activity Following Injury: Towards Understanding a More Accessible Solution for Shorter Recovery Time.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Farag Hanafy, Lecturer of Biomechanics, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Cryotherapy and Balance
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Cryotherapy
Keywords: Postural Stability; Public Health; Balance
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into one of two locations of the cryotherapy application. Some began the session with cryotherapy being applied on their ankle evertors, while others began the session with the cryotherapy being applied on their hip adductors.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle evertors (Active Comparator): Ice packs will be applied to the selected muscles according to the random selection that will be performed previously. The ice bags will be filled with crushed ice, weighing approximately one half of a kilogram. They will be wrapped in a thin cotton towel, and applied on the skin along the anatomical location of the tested muscles. For the ankle evertors, the ice bag will be applied to the lateral side of the ankle encompassing the lateral malleolus.The cryotherapy session will be lasted for exactly 20 minutes . Sessions will be separated by a 30-minute rest interval
  Interventions: Other: Cryotherapy
- Hip adductors (Active Comparator): Ice packs will be applied to the selected muscles according to the random selection that will be performed previously. The ice bags will be filled with crushed ice, weighing approximately one half of a kilogram. They will be wrapped in a thin cotton towel, and applied on the skin along the anatomical location of the tested muscles. For the hip adductors, the ice bag will be applied to the medial side of the thigh, covering the entire area from the groin, to just above the knee joint. The cryotherapy session will be lasted for exactly 20 minutes . Sessions will be separated by a 30-minute rest interval
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — Crushed ice in a plastic bag will be used, as it is a widely accessible and financially convenient method of cryotherapy. One half of a kilogram of ice will be placed in a plastic bag. The plastic bags will be 17 cm wide and 22 cm long. The air will be squeezed out of the bag and it will be sealed. The bag will be wrapped in a wet towel and applied to the tested area. Every five bags of crushed ice will be kept in an insulated foam container containing one kilogram of dry ice. Dry ice has a temperature of negative 80 degrees Celsius, and is used to keep the bags of crushed ice in a frozen state till the participants are briefed and the testing began.

SUMMARY:
The purpose of this study is to investigate the effect of cryotherapy application on hip adductors and ankle evertors on the Overall Stability Index (OSI), the Medio-Lateral Stability Index (MLSI), and the Antero-Posterior Stability Index (APSI) in healthy adult females.

DETAILED DESCRIPTION:
Cryotherapy is one of the most common and inexpensive forms of treatment for both acute and chronic injuries. Yet, there is a deficiency in research concerning the impact of cooling on balance in healthy females

ELIGIBILITY:
Inclusion Criteria:

* healthy females will participate in this study. All participants should have unrestricted ankle and hip joints range of motion as well as ankle and hip muscles strength grade four to five (using manual muscle testing).

Exclusion Criteria:

* Participants will be excluded from the study if they had any previous history of hip or ankle joint neuromuscular or musculoskeletal injury or surgery, any pathology to the hip or ankle joints (i.e. abnormal ligament laxity and congenital deformities), any problems related to balance and stability.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Stability Index | changes from Baseline to immediately after the cryotherapy application
  The Stability Index represented the variance of platform displacement in degrees from a leveled position in both the AP and ML directions. A high number is indicative of poor neuromuscular control, which may increase the potential for orthopedic injury or falling.

SECONDARY OUTCOMES:
Medio-lateral Postural Stability Index | changes from Baseline to immediately after the cryotherapy application
Antero-posterior Postural Stability index | changes from Baseline to immediately after the cryotherapy application

CONTACTS AND LOCATIONS:
Overall Officials: Ayman G Matar, PhD, Study Director — Lecturer of Biomechanics; Nagui S Nassif, Prof., Study Chair — Assistant Professor of Biomechanics; Naglaa M Elhafez, Prof., Study Chair — Professor of Biomechanics; Ghada M Elhafez, Prof., Study Director — Professor of Biomechanics; Sondus Hassounah, Public Health Teaching Fellow, Study Chair — Public Health Teaching Fellow

REFERENCES:
- [Background] Algafly AA, George KP. The effect of cryotherapy on nerve conduction velocity, pain threshold and pain tolerance. Br J Sports Med. 2007 Jun;41(6):365-9; discussion 369. doi: 10.1136/bjsm.2006.031237. Epub 2007 Jan 15. PMID 17224445
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753